CLINICAL TRIAL: NCT00817505
Title: A Randomized, Open, Single-Dose, Single-Centre, Cross-over, Phase I Study in Type 1 Diabetes Mellitus Patients to Estimate the Extent and Rate of Absorption of AZD1656 After Administration of a Tablet Formulation in the Fasting State and Just Before Food in Comparison With an Oral Suspension of AZD1
Brief Title: To Evaluate the Bioavailability of a Tablet of AZD1656
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Klas Malmberg, MD, PhD, Prof. Medical Science Director, Emerging Products, AstraZeneca Pharmaceuticals
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: D1020C00010
Record Dates: First submitted 2008-12-24; First posted 2009-01-06 (Estimated); Last update posted 2009-11-03 (Estimated); Status verified 2009-11

CONDITIONS: Type 1 Diabetes
Keywords: Type I diabetes; bioavailability
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — AZD1656

ARMS (3):
- 1 (Active Comparator): AZD1656 tablet + food
  Interventions: Drug: AZD1656
- 2 (Active Comparator): AZD1656 susp. without food
  Interventions: Drug: AZD1656
- 3 (Active Comparator): AZD1656 tablet
  Interventions: Drug: AZD1656

INTERVENTIONS:
Drug: AZD1656 — Single dose oral tablet
Drug: AZD1656 — Single dose oral suspension

SUMMARY:
To evaluate the bioavailability of a tablet of AZD1656.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, type I diabetes patients, female with non child-bearing potential.
* Treated with insulin for more than 3 years. Well controlled HbA1c.
* Have a body mass index (BMI) ≥19 and ≤35

Exclusion Criteria:

* Clinically significant illness except type I diabetes, or clinically relevant trauma, as judged by the investigator, within 2 weeks before the first administration of the investigational product
* Daily use of nicotine containing substances.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2008-12; Primary Completion 2009-03 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic variables ( Area under the plasma concentration vs. time curve (AUC), maximum plasma concentration (Cmax), time to reach maximum plasma concentration (tmax), terminal elimination half-life (t½) and apparent oral clearance (CL/F) | Blood samples taken up to 72 hours

SECONDARY OUTCOMES:
Pharmacodynamic variables (Plasma glucose) | Taken repeatedly during treatment periods
Safety Variables (AEs, BP, pulse, electrocardiogram (ECG), hypoglycaemic symptoms and laboratory variables) | Taken during treatment periods

CONTACTS AND LOCATIONS:
Overall Officials: Klas Malmberg, MD, PhD, Prof, Study Director — AstraZeneca R&D Mölndal; Emanuel P DeNoia, MD, Principal Investigator — Healthcare Discoveries LLC Icon Development Solutions
Locations (1):
- Research site, San Antonio, Texas, United States